CLINICAL TRIAL: NCT02342379
Title: A Phase 2, Investigator Initiated Study to Determine the Safety and Efficacy of TH-302 in Combination With Bevacizumab for Glioblastoma Following Bevacizumab Failure
Brief Title: TH-302 in Combination With Bevacizumab for Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRC 12-0105; HSC20130212H (Other: UT Health Science Center Institutional Review Board)
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and TH-302 (Experimental): Patients will be treated with combination of bevacizumab and TH-302.
  Interventions: Drug: Bevacizumab; Drug: TH-302

INTERVENTIONS:
Drug: Bevacizumab — 10mg/kg
  Other Names: Avastin
Drug: TH-302 — 670mg/m2
  Other Names: MSC2491899A

SUMMARY:
Dual center, single arm, two-stage, non-blinded, prospective study of combination therapy bevacizumab at 10mg/kg and TH-302 at 670mg/m2 every 2 weeks (6 week cycle) until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Histologically confirmed glioblastoma
* Progression following both standard combined modality treatment with radiation and temozolomide chemotherapy, as well as bevacizumab
* Recovered from toxicities of prior therapy to grade 0 or 1
* ECOG performance status ≤ 2
* Life expectancy of at least 3 months
* Acceptable liver function:

  1. Bilirubin ≤ 1.5 times upper limit of normal
  2. AST (SGOT) and ALT (SGPT) ≤ 3.0 times upper limit of normal (ULN);
* Acceptable renal function:

  a. Serum creatinine ≤ULN
* Acceptable hematologic status (without hematologic support):

  1. ANC ≥1500 cells/uL
  2. Platelet count ≥100,000/uL
  3. Hemoglobin ≥9.0 g/dL
* All women of childbearing potential must have a negative serum pregnancy test and male and female subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose

Exclusion Criteria:

* The subject is receiving warfarin (or other coumarin derivatives) and is unable to switch to low molecular weight heparin (LMWH) before the first dose of study drug.
* The subject has evidence of acute intracranial or intratumoral hemorrhage either by MRI or computerized tomography (CT) scan. Subjects with resolving hemorrhage, punctate hemorrhage, or hemosiderin are eligible.
* The subject is unable to undergo MRI scan (eg, has pacemaker).
* The subject has received enzyme-inducing anti-epileptic agents within 14 days of study drug (eg, carbamazepine, phenytoin, phenobarbital, primidone).
* The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 Grade ≤ 1 from AEs (except alopecia, anemia and lymphopenia) due to surgery, antineoplastic agents, investigational drugs, or other medications that were administered prior to study drug.
* The subject has evidence of wound dehiscence
* Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause normal tissue hypoxia
* The subject is pregnant or breast-feeding.
* The subject has serious intercurrent illness, such as:

  1. hypertension (two or more blood pressure [BP] readings performed at screening of > 150 mmHg systolic or > 100 mmHg diastolic) despite optimal treatment
  2. non-healing wound, ulcer, or bone fracture
  3. significant cardiac arrhythmias
  4. untreated hypothyroidism
  5. uncontrolled active infection
  6. symptomatic congestive heart failure or unstable angina pectoris within 3 months prior study drug
  7. myocardial infarction, stroke, transient ischemic attack within 6 months
  8. gastrointestinal perforation, abdominal fistula, intra- abdominal abscess within 1 year
  9. history or clinical evidence of pancreatitis within 2 years
* The subject has inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* The subject has received any of the following prior anticancer therapy:

  1. Non-standard radiation therapy such as brachytherapy, systemic radioisotope therapy, or intra-operative radiotherapy (IORT). Note: stereotactic radiosurgery (SRS) is allowed
  2. Non-bevacizumab systemic therapy (including investigational agents and small-molecule kinase inhibitors) or non-cytotoxic hormonal therapy (eg, tamoxifen) within 7 days or 5 half-lives, whichever is shorter, prior first dose of study drug
  3. Biologic agents (antibodies, immune modulators, vaccines, cytokines) within 21 days prior to first dose of study drug
  4. Nitrosoureas or mitomycin C within 42 days, or metronomic/protracted low-dose chemotherapy within 14 days, or other cytotoxic chemotherapy within 28 days, prior to first dose of study drug
  5. Prior treatment with carmustine wafers
  6. Prior treatment with TH-302

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-05; Primary Completion 2019-01-04 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brenner, MD, Principal Investigator — University of Texas Health Science Center San Antonio at the Cancer Therapy and Research Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Texas Health Science Center San Antonio at the Cancer Therapy and Research Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab and TH-302
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and TH-302
Number analyzed (Participants) | 35
Age, Customized [Count of Participants; unit: Participants]
  18-21 years | 1
  22-29 years | 4
  30-39 years | 7
  40-49 years | 4
  50-59 years | 11
  60-69 years | 6
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White : Female | 10
  White : Male | 15
  Black or African American : Female | 0
  Black or African American : Male | 1
  White/Hispanic or Latino : Female | 1
  White/Hispanic or Latino : Male | 6
  Asian : Female | 0
  Asian : Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: Safety lab tests and adverse event assessment
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab and TH-302
Number analyzed (Participants) | 35
Participants | 35

2. Secondary Outcome: Progression Free Survival
Description: Progression of disease by RANO criteria:
  The RANO criteria divides response into four types of response based on imaging and clinical features
  1. complete response
  2. partial response
  3. stable disease
  4. progression
Time Frame: 4 months
Population: 3 of the enrolled participants were not evaluable
Measure: Number; unit: Number of participants
Arm/Group | Bevacizumab and TH-302
Number analyzed (Participants) | 32
Number of participants | 32

ADVERSE EVENTS:
Time Frame: Adverse events are collected from start of drug administration until 30 days after study drug is discontinued, giving a total of 5 months potential evaluation period.
Arm/Group | Bevacizumab and TH-302
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 35/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and TH-302 (N=35)
Abscess (left axillary abscess) (Skin and subcutaneous tissue disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 3 (6)
Anorexia (Gastrointestinal disorders) | 1 (1)
Cognitive Disturbance (Nervous system disorders) | 1 (1)
confusion (Nervous system disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Decreased Appetite (Gastrointestinal disorders) | 2 (2)
Decreased Platelets (Blood and lymphatic system disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Edema (pedal) (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (intermittent) (Vascular disorders) | 1 (1) — Bleeding of the nose
Facial Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Blurred vision/diplopia (Eye disorders) | 2 (2)
Fatigue (General disorders) | 12 (13)
Fever (General disorders) | 1 (2)
Flu (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Upper respiratory tract infection
Headache (Nervous system disorders) | 2 (3)
Heartburn (Gastrointestinal disorders) | 1 (1)
Hemorrhoid (Skin and subcutaneous tissue disorders) | 2 (2)
Herpes Simplex Virus (Infections and infestations) | 1 (1)
Hoarsness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) — palmar plantar erythrodysethesia syndrome
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 (6)
Hypertension (Cardiac disorders) | 2 (3) — High blood pressure
Kratoderma (Skin and subcutaneous tissue disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) — Decreased white blood cell count
Lung Infection (PNA) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mouth Sores (Gastrointestinal disorders) | 1 (1)
Anal Mucositis (Skin and subcutaneous tissue disorders) | 6 (7)
Oral Mucositis (Gastrointestinal disorders) | 5 (9)
Perianal Mucositis (Skin and subcutaneous tissue disorders) | 3 (6)
Rectal Mucositis (Gastrointestinal disorders) | 2 (2)
Vaginal Mucositis (Reproductive system and breast disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9)
Neutropenia (Blood and lymphatic system disorders) | 4 (9)
Pain, abdominal (Gastrointestinal disorders) | 2 (2)
Pain, rectal (Gastrointestinal disorders) | 2 (2)
Phlebitis (Blood and lymphatic system disorders) | 1 (1) — Left anticubital fossa
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Proteinuria (Endocrine disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 9 (11)
Scar (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Abrasion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1 (1) — Peeling
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) — Groin
Skin excoriation (Skin and subcutaneous tissue disorders) | 1 (1) — Right armpit
Other skin excoriation (Skin and subcutaneous tissue disorders) | 1 (2) — Labial/vaginal/rectal
Skin Ulceration (Skin and subcutaneous tissue disorders) | 6 (9)
Small intestine perforation (Gastrointestinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (19)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 2 (3)
Vaginal Infection (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Weakness (General disorders) | 1 (1) — Left sided weakness
Wound complication (Skin and subcutaneous tissue disorders) | 1 (1) — Delayed healing of right chest wall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT02342379/Prot_SAP_000.pdf